CLINICAL TRIAL: NCT05191654
Title: Investigation of Cardiopulmonary Parameters, Motor Development and Muscle Strength in Children With Down Syndrome With and Without Congenital Heart Disease
Brief Title: Investigation of Cardiopulmonary Parameters, Motor Development and Muscle Strength in DS With and Without CHD
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Tuğba Şanlı, Principal Investigator, Atılım University
Other Study IDs: 59394181-604.01.01-75
Record Dates: First submitted 2021-10-27; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Congenital Heart Defects; Down Syndrome; Gross Motor Development Delay
Keywords: congenital heart defects; Down syndrome; motor skills
MeSH Terms: conditions — Heart Defects, Congenital; Down Syndrome | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with Congenital heart diseases
  Interventions: Diagnostic Test: evaluation of cardiopulmonary parameters, gross motor development and hand grip strength
- without Congenital heart diseases
  Interventions: Diagnostic Test: evaluation of cardiopulmonary parameters, gross motor development and hand grip strength

INTERVENTIONS:
Diagnostic Test: evaluation of cardiopulmonary parameters, gross motor development and hand grip strength — Gross motor development was evaluated with Gross Motor Function Measure (GMFM-88). Hand grip strength was measured with the Baseline Pneumatic Bulb Dynamometer. Cardiopulmonary parameters values was evaluated with echocardiography.

SUMMARY:
Congenital heart diseases (CHD) are detected in 40-60% of individuals with Down syndrome (DS) and increase the risk of developmental delay in the presence of syndromes. The aim of the study was to compare cardiopulmonary parameters, gross motor development and hand grip strength in DS children with and without CHD. Demographic variables, cardiopulmonary parameters and echocardiographic values were recorded. Gross motor development was evaluated with Gross Motor Function Measure (GMFM-88). Hand grip strength was measured with the Baseline Pneumatic Bulb Dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Down syndrome as a result of genetic analysis,
* For the congenital heart disease group; undergoing cardiac surgery at least 6 months before the evaluation, diagnosed as CHD by a pediatric cardiologist based on echocardiographic findings,
* For the group without congenital heart disease, patients who have not undergone cardiac surgery, are asymptomatic with a septal defect smaller than 4-5 mm, are expected to close, and are hemodynamically normal by a pediatric cardiologist,
* Children whose families were informed about the study and gave written consent to participate in the study were included in the study.

Exclusion Criteria:

* Having another genetic abnormality other than Down syndrome,
* undergoing surgery other than cardiac surgery,
* Having an orthopedic or neurological problem,
* Respiratory support,
* With atlantoaxial instability,
* Children with hematological disease were not included in the study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with down syndrome
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 | october 2020- june 2021
  Gross motor development of the participants was evaluated with the Gross Motor Function Measure-88 questionnaire. The value as a percentage was obtained as a result of the survey. Gross Motor Function Measure-88 consists of 5 sections that include the evaluation of Lying & Rolling, Sitting, Crawling & Kneeling, Standing, Walking, Running & Jumping activities. Each item in the sections consists of a 4-point scale. Scores for each section are summed and divided by 5.The maximum score on the scale is 100. A high score indicates good gross motor development.
  0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes
Bulb Dynamometer | october 2020- june 2021
  Hand grip strength was measured with a Baseline Pneumatic Bulb Dynamometer (Fabrication Enterprises INC, Elmsford, NY USA). With a bulb dynamometer, the spherical grip force is measured using a rubber balloon tip. The bulb dynamometer has 3 removable sizes. The values measured on the manometer are recorded in kPa. The measurement is repeated 3 times and the highest value is taken.
Left ventricular ejection fraction (EF) | october 2020- june 2021
  Echocardiographic findings performed in the last 6 months were evaluated by a pediatric cardiologist. It is obtained by dividing the difference in left ventricular volume at end-diastolic and end-systolic by the end-diastolic left ventricular volume. Left ventricular ejection fraction (EF) indicate the systolic function of the left ventricle. Ejection fraction value show as a percentage (%). The ejection fraction normal value is between 50 percent and 70 percent.
Interventricular septum wall thickness (IVS) | october 2020- june 2021
  Echocardiographic findings performed in the last 6 months were evaluated by a pediatric cardiologist. It is important in the risk classification potential of left ventricular systolic function. Its value is show as millimeters (mm).
Left ventricular end-diastolic diameter (LVDd) | october 2020- june 2021
  Echocardiographic findings performed in the last 6 months were evaluated by a pediatric cardiologist. It is important in the risk classification potential of left ventricular systolic function. Its value is show as millimeters (mm).
Fractional shortening (FS) | october 2020- june 2021
  Echocardiographic findings performed in the last 6 months were evaluated by a pediatric cardiologist. Fractional shortening evaluates left ventricular systolic function. Fractional shortening value show as a percentage (%). The value of normal fractional shortening in children is between 28-44%.
Wang Respiratory Score | october 2020- june 2021
  The Wang respiratory score assesses respiratory frequency, wheezing, retraction, and general condition. parameters are scored between 0-3 and summed. A higher score indicates that the situation is getting severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No